CLINICAL TRIAL: NCT03147625
Title: Salutogenic Healthy Aging Program Embracement (SHAPE) for Elderly-only Households
Acronym: SHAPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Boon Lay Constituency (Unknown); Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Wang Wenru, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOE-SSTRG
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Elderly
Keywords: Aged; Independent living; Health Promotion; Residence Characteristics; Elderly-only household

STUDY DESIGN:
Intervention Model Description: In this two-armed randomized controlled trial, participants will be allocated to either the intervention group or the control group through stratified permuted block randomization. Participants in the intervention will undergo SHAPE while participants assigned to the control group will receive usual care, which refers to existing community services provided by the local community centre, senior activity centre and voluntary welfare organisations.
Who Masked: Outcomes Assessor
Masking Description: A research nurse not involved in the delivery of SHAPE intervention will be blinded to the participants' group assignment to conduct data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHAPE Intervention (Experimental): Participants in this group will receive a 12-week SHAPE intervention, comprising of 2 home visits, 10 weekly group-based activity sessions and a SHAPE health-promotion booklet.
  Interventions: Behavioral: SHAPE Intervention
- Control group (No Intervention): Participants in the control group will continue to participate in activities offered in the senior activity centre, community centres and voluntary welfare organisations.

INTERVENTIONS:
Behavioral: SHAPE Intervention — SHAPE seeks to identify, equip and strengthen resources in elderly residing in elderly-only households. The content will be further developed according to the findings of an existing descriptive qualitative study, literature review and a multi-disciplinary expert panel review. The home visit will involve assessment, observation and evaluation of elderly' health status, lifestyle and home environment, followed by guidance on health-promoting behaviour and emphasis on strengthening inner health resources. This provides an individualized approach to enhance personal health skills. Group-based activity sessions are directed to facilitate group interaction among peers as well as equipping and enhancing external resources.
  Arms: SHAPE Intervention

SUMMARY:
Elderly residing in elderly-only households are more vulnerable as they are socially isolated, suffer from poorer health outcomes, and are less likely to adopt health-promoting behaviors. While multi-dimensional preventive home visits provide older adults with the individualized care to cope with living in their homes, group-based education promotes peer learning and allows for social interaction. Elderly residing in elderly-only households can reap the benefits derived from the coaction of preventive home visits and group-based education, providing them with the personalized care to age healthily in their homes and a platform to develop social connectedness with their peers. This study uses the combination of preventive home visit and group-based education program to promote healthy aging in elderly living in elderly-only households.

Using a randomized controlled trial, the study aims to evaluate the effectiveness of a 12-week health promotion and risk prevention program, named Salutogenic Healthy Aging Program Embracement (SHAPE) for elderly-only households. Participants in the experimental group will receive 2 home visits, 10-weekly group-based activity sessions and a SHAPE health-promotion booklet. A process evaluation using face-to-face interviews will also be conducted for elderly receiving SHAPE to explore their views on the program.

The use of salutogenic model breaks away from the negatively connoted conventional biomedical model and addresses on optimization of positive health. Ultimately, the SHAPE intervention seeks to identify, equip and strengthen resources for elderly-only households, encouraging the adaption of health-promoting and risk-preventing actions to achieve better health outcomes and higher quality of life.

DETAILED DESCRIPTION:
Aim and Hypothesis This study aims to develop and evaluate the effectiveness of a multi-dimensional, community-based health promotion and prevention program, SHAPE, on sense of coherence, self-efficacy, quality of life, health-promoting behaviours, and health-related outcomes among elderly residing in elderly-only households in Singapore.

It is hypothesized that compared with participants in the control group, participants in the experimental group will have improved sense of coherence, better quality of life, increase uptake of health-promoting behaviours, higher self-efficacy and other health outcomes.

Study Design A single-blinded two-arm, randomized controlled trial (RCT), pretest and repeated post-test design will be used. The study will be conducted in a small residential estate located in the west of Singapore. Stratified permuted block randomization will be used to allocate participants into experimental and control group. The 12-week SHAPE will be provided to elderly living in the blocks allocated to the experimental group, and both groups will receive usual activities offered in senior activity centre, community centre and voluntary welfare organisations. One research nurse (RN) together with a research assistant A (RA A) who has social work background will conduct the intervention, and another research assistant B (RA B) will conduct the data collection. The RA B will be blinded to participants' group assignment to prevent subjective bias stemming from the knowledge of grouping. Four measurements will be conducted at baseline prior to the intervention, at 3 months immediately after the intervention, 6 months, and 12 months from the baseline.

Sample Size Power analysis calculation on sample size is based on previous studies on community-based programs conducted in community-dwelling older adults which reported sense of coherence having a medium effect size (d=0.46-0.57). Sample size calculation is therefore calculated based on a medium effect size of 0.5. A minimum sample size of 64 participants in each group is needed to detect a difference between groups at an alpha of 0.05 and power of 0.80. We estimate 20% attrition rate, a total of 154 participants would be needed, with 77 in each group

Randomization To account for differences in living arrangement and ensure that elderly living in the same household are assigned to the same intervention or control group, stratified permuted block randomization will be used in this study. Participants will be grouped according to either of the three strata: (1) single elderly in a household, (2) two elderly from same household participating in the trial (a pair) and (3) only one out of two elderly from same household participating in the trial. Blocks of 10, with the assignment of 5 to experimental group and 5 to control group, will be used for each strata. Using a computerized randomization software, a statistician will generate the randomization list and prepare 3 different sets of sealed envelopes. According to their strata, the participant or the pair of participants will choose from the respective set of envelopes themselves to determine the group assignment.

Intervention Group A 12-week SHAPE intervention, comprising of 2 home visits, 10 weekly group-based activity sessions and a SHAPE health-promotion booklet, is proposed.

SHAPE seeks to identify, equip and strengthen resources for elderly residing in elderly-only households. The content of program will be further developed and mould by the results from an existing qualitative study, literature review and by a group of multi-disciplinary expert panel consisting of gerontology-trained nurses, physiotherapist, occupational therapists and social workers and well-established researchers. Homes visits and group-based activity sessions will be conducted by the researchers, who are a trained RN and a trained RA A with social work background The home visit will involve assessment, observation and evaluation of elderly' health status, lifestyle and home environment, followed by guidance on health-promoting behaviour and emphasis on strengthening inner health resources. This will provide an individualized approach to enhance personal health skills. Group-based activity sessions are directed to facilitate group interaction among peers as well as equipping and enhancing external resources to the older adults. Homework will be given at the end of each session to allow them to reflect on the contents of each session. Special considerations will be taken during the design of SHAPE health-promotion booklet to cater to older people's needs such as larger prints, shorter sentences and pictorial examples. Two voluntary older adults will also be involved in shaping the content of the booklet.

Control Group/Usual Care:

Participants in the control group will continue to participate in activities offered in senior activity centres, community centres and voluntary welfare organisations.

Outcome Measures Sense of coherence, quality of life, self-rated health, health-promoting behaviors, self-efficacy, functional mobility, instrumental activities of daily living, body mass index, blood pressure, fasting blood glucose, cognitive function, depressive symptoms, anxiety, perceived stress, social support, hospital admissions

Semi-structured Interviews: Process Evaluation To explore the responsiveness, strengths and weaknesses of SHAPE, a qualitative face-to-face interview will be conducted after the start of intervention at 6 months. Purposive sampling will be used and participants from the experimental group will be interviewed. A semi-structured interview guide will be used to explore the perspectives of participants towards the responsiveness and usefulness of SHAPE, as well as to understand the strengths and weaknesses of the program and identify areas for future improvement. All interviews will be conducted by the researcher till data saturation.

Data Collection Upon the approval of ethics, the researcher will collaborate with the site-PI from the community and volunteers from residents' committee to recruit study participants. Eligibility of participants will be assessed face-to-face by researcher nurse before obtaining informed consent. Data on socio-demographics, past medical history and health conditions will also be collected. Data will be collected at 4 different intervals: baseline (pre-test), 3 months (post-test 1), 6 months (post-test 2) and 12 months (post-test 3) from the baseline. The RA B will arrange appointment with participants to collect the data through face-to-face interview as some older adults might be illiterate and are unable to self-administer the questionnaire.

Data Analysis Data will be analysed using SPSS version 24. Baseline categorical demographic characteristics between the experimental and control groups will be examined using Chi-squared or Fisher's Exact test. Independent t-test will be used for quantitative variables if normality and homogeneity assumptions are satisfied; otherwise Mann-Whitney U-test will be used. Repeated measures analysis of variance (ANOVA) will be performed to analyse the interaction effect (time x group) between two groups on numerical outcomes over time, setting level of significance at p<0.05 for two-tailed test. In addition, General Linear Mixed Model (GLM) will be used to compare the study outcomes between two groups at each time point. To correct for type 1 error on multiple comparisons for each time point, statistical significance will be set at p < 0.01.

Qualitative thematic analysis will be used to analyse the data collected from the interviews. All interviews are audio-taped. Interviews will be conducted and transcribed in either in Chinese or English language respectively. Co-researcher will check for any discrepancy between the English and Chinese transcripts to ensure the congruency of meaning in data.

Potential impact The SHAPE intervention aims to equip older adults living alone with both internal and external resources and encourage the adaption of health-promoting and risk-preventing behaviours to promote healthy aging. Targeting on the group of vulnerable and poorer older population, the program seeks to optimize health by enhancing one's ability to cope with health and age-related stressors and promote independent living, preventing functional dependence.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling elderly aged 65 years and above,
* either living by himself/herself or living his/her older spouse or living with an unrelated elderly
* able to comprehend and converse either in English or Chinese language
* able to be followed up on home visits.

Exclusion Criteria:

Elderly who

* have significant cognitive impairment (Mini Mental State ≤ 23)
* have severe hearing and/or visual impairment
* have terminal illness with life expectancy <12 months
* have uncontrolled psychiatric disorders
* are on home visit follow-ups with other organizations
* are involved in existing clinical trials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Sense of Coherence | Baseline, 3 months, 6 months, 12 months
  Sense of coherence refers to one's ability to comprehend, make sense of and mobilize resources to cope with stressors. The 13-item Orientation to Life Questionnaire (SOC-13) measuring sense of coherence consists of 3 domains: comprehensibility (5-item), manageability (4-item) and meaningfulness (4-item). The higher the score, the better the sense of coherence.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, 3 months, 6 months, 12 months
  The World Health Organisation Quality of Life- Older Adults questionnaire (WHOQoL-OLD) is a 24-item valid and reliable cross-cultural geriatric-centric instrument consisting of 6 subscales: sensory abilities, autonomy, past, present and future, social participation, death and dying and intimacy. The total score ranges from 24 to 120, with higher scores suggesting higher quality of life.
Change in Self-rated Health | Baseline, 3 months, 6 months, 12 months
  Participants will be asked to rate their own health on both the self-rated health likert-scale item, as well as the self-rated health visual analogue scale from EQ-5D instrument (range 0 to 100).
Change in Health-Promoting behaviors | Baseline, 3 months, 6 months, 12 months
  The Health promotion lifestyle profile-II (HPLP-II) is an established instrument measuring multi-components of health promotion lifestyle behaviors.It uses 4-point likert scale (4-routinely to 1-never) to reflect how often the individual engages in the listed health-promoting behavior. The total score ranges from 30 to 120, with higher scores suggesting greater engagement in health promoting behaviors.
Change in Self-efficacy | Baseline, 3 months, 6 months, 12 months
  The Generalised Self-efficacy Scale (GSE) was developed to assess perceived self-efficacy with the intention to predict coping with daily events and adaptation of stressful life events. It has 10 items and they are rated on a 4-point likert scale. A higher score indicates better ability to cope with stressful situations.
Change in Instrumental Activities of Daily Living | Baseline, 12 months
  The Lawton's Instrument Activities of Daily Living (IADLs) instrument is used to assess one's independent living skills. Higher total scores portray higher independence and functional ability of an individual
Change in Functional Mobility | Baseline, 3 months, 6 months, 12 months
  The Time-Up Go test (TUGT) is a simple, quick and widely used clinical test to assess lower extremity function, mobility and fall risk, even in healthy older adults. Participants will be asked to stand up from a standard chair, walk a distance of three metres, turn, walk back and sit down. While routine walking aids are allowed, they are not permitted to use their arms to stand up and no physical assistance is offered. A stopwatch will be used to record the time to complete the task and the average time of 2 attempts will be taken as a reading. Shorter times reflect better functional mobility.
Change in Blood Pressure | Baseline, 3 months, 6 months, 12 months
  Participants are to rest and stabilize for 10 minutes before taking their systolic and diastolic using a standard mercury sphygmomanometer on the right upper arm (unless contraindicated)
Change in Fasting Blood glucose | Baseline, 3 months, 6 months, 12 months
  Participants will be asked to fast for at least 6 hours prior to test for fasting blood glucose. A standardized glucometer will be used to determine the reading of fasting blood glucose.
Change in Body Mass Index | Baseline, 3 months, 6 months, 12 months
  A standardised weighing machine and measuring tape will be used to measure the height and weight of the participant.
Change in Cognitive function | Baseline, 12 months
  The Mini Mental State Examination (MMSE) is used to assess and detect for any cognitive impairment. The summed scores of MMSE range from 0-30. The higher the score, the better the cognitive function.
Change in Depressive Symptoms | Baseline, 3 months, 6 months, 12 months
  The 15-item Geriatric Depression scale (GDS) was developed to screen for depressive symptoms in older adults and is a well-validated depression screening tool used in Singapore. Its total score range from 0 to 15. The higher the score, the higher one presents with depressive symptoms.
Change in Anxiety | Baseline, 3 months, 6 months, 12 months
  The 20-item Geriatric Anxiety Inventory (GAI) measures common typical anxiety symptoms in older adults. Its total score ranges from 0 to 20; higher summed scores refers to higher anxiety levels.
Change in Perceived Stress | Baseline, 3 months, 6 months, 12 months
  The 10-item Perceived Stress Scale (PSS) will be used to assess subjective stress levels in individuals. Its total range from 0 to 40, and higher scores denotes higher perceived stress.
Change in Perceived Social Support | Baseline, 3 months, 6 months, 12 months
  The Duke Social Support Index (DSSI) will be used to assess subjective social support among elderly. The abbreviated version (DSSI-10) consists of 10 items, each on a 3-point likert scale, and measures the following two constructs: social interaction and social satisfaction. Possible score ranges from 10 to 30 and higher scores reflect higher levels of perceived support support.
Change in Hospital admissions | Baseline, 12 months
  Frequency of hospital admissions in the past 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wenru Wang, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Seah B, Espnes GA, Hong WT, Wang W. Salutogenic Healthy Ageing Programme Embracement (SHAPE)- an upstream health resource intervention for older adults living alone and with their spouses only: complex intervention development and pilot randomized controlled trial. BMC Geriatr. 2022 Dec 3;22(1):932. doi: 10.1186/s12877-022-03605-3. PMID 36460959